CLINICAL TRIAL: NCT07278739
Title: A Randomized Controlled Trial of an Intervention Called "Algorithm-Enabled Patients Activated in Cancer Care Through Teams" (A-PACT) to Improve Goals of Care Communication for People With Cancer
Brief Title: Testing an Educational Program to Improve Goals of Care Conversations Between Patients and Their Care Teams
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S2424CD; NCI-2025-08258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2424CD (Other: SWOG); SWOG-S2424CD (Other: DCP); S2424CD (Other: CTEP); R37CA296075 (NIH); UG1CA189974 (NIH)
Record Dates: First submitted 2025-12-05; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Randomization assignment is not revealed to clinicians and general staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Usual care + A-PACT) (Experimental): Patients attend an initial A-PACT education session over 30-45 minutes by phone and receive follow-up A-PACT phone calls over 15 minutes each twice monthly, or less frequently per patient preference, for up to 6 months, in addition to usual care.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Interview; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention
- Group 2 (Usual care) (Active Comparator): Patients receive usual care for 6 months.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive A-PACT education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group 1 (Usual care + A-PACT)
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
  Arms: Group 1 (Usual care + A-PACT)
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive A-PACT phone calls
  Arms: Group 1 (Usual care + A-PACT)

SUMMARY:
This clinical trial evaluates an educational program called Algorithm-Enabled Patients Activated in Cancer Care Through Teams (A-PACT) for reducing unplanned hospital visits and improving goals of care conversations with providers among patients with solid cancers. A-PACT is an educational program where lay health workers (educators) help patients talk with their health care team about issues that matter most to them (goals of care). During A-PACT sessions, patients receive assistance in formulating health care and end of life care preferences, assistance in completing advance directives, guidance on how to engage in these conversations with family members, friends, and clinical teams, and encouragement to discuss these topics with their clinical team. A-PACT may reduce unplanned hospital visits and improve goals of care communication with providers among patients with solid cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the proportion of participants who have any hospitalizations within 12 months after randomization between those receiving A-PACT (intervention arm) and those receiving usual care alone (control arm).

SECONDARY OBJECTIVES:

I. To compare the proportion of participants who report anxiety at 3 months compared to baseline between participants receiving A-PACT and participants receiving usual care.

II. To compare the proportion of participants who report depression at 3 months compared to baseline between participants receiving A-PACT and participants receiving usual care.

III. To assess the proportion of participants who receive intensive end-of-life care between participants receiving A-PACT and those receiving usual care alone.

IMPLEMENTATION OBJECTIVES:

I. To quantitatively and qualitatively assess how patient, clinician, and organizational factors shape effectiveness and implementation of A-PACT.

II. To measure feasibility of machine learning (ML) algorithm, adoption of intervention (patient enrollment), and fidelity (% of patients completing A-PACT).

EXPLORATORY OBJECTIVES:

I. To assess the following in participants on the intervention arm versus the usual practice arm:

Ia. The proportion of participants who have any hospitalization or emergency department visits within 12 months from randomization between those receiving A-PACT and those receiving usual care; Ib. The mean number of hospitalizations within 12 months from randomization between participants receiving A-PACT and participants receiving usual care alone; Ic. The mean number of hospitalizations or emergency department visits within 12 months of randomization between participants receiving A-PACT and participants receiving usual care alone; Id. Anxiety at 6 months from baseline; Ie. Depression at 6 months from baseline; If. Heard and Understood measures at 6 months from baseline; Ig. Prognostic awareness and treatment preferences at 6 months from baseline; Ih. Presence of goals of care documentation in the electronic health record at 12 months; Ii. Presence of advance directive documentation in the electronic health record at 12 months; Ij. Presence of physician orders for life sustaining treatment documentation in the electronic health record at 12 months; Ik. The potential differential impact of sociodemographic factors on all outcomes.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 1: Patients attend an initial A-PACT education session over 30-45 minutes by phone and receive follow-up A-PACT phone calls over 15 minutes each twice monthly, or less frequently per patient preference, for up to 6 months, in addition to usual care.

GROUP 2: Patients receive usual care for 6 months.

After completion of study intervention, patients are followed up at months 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of a solid tumor malignancy of any stage
* Participants must be identified as high risk, defined as having 6 month mortality estimate from machine learning (ML) algorithm >= 20%
* Participants must not be receiving or have pre-existing plans to enter hospice care at the time of study registration
* Participant must be actively receiving or planning to receive systemic anti-cancer therapy (defined as any oral, injection, or intravenous therapy against cancer) within 3 months after registration

  * NOTE: This includes chemotherapy (conventional or cytotoxic chemotherapy), hormone therapy, targeted therapy, and immunotherapy
  * NOTE: Participants are allowed to be co-enrolled on other clinical trials including trials using investigational agents
* Participants must be >= 18 years of age at the time of study enrollment
* Participants who can complete Patient Reported Outcome (PRO) questionnaires in English or Spanish must be willing to 1) complete PROs at all scheduled assessments; and 2) complete the pre-registration (baseline) PRO forms within 14 days prior to registration
* Participants must be able to provide a valid telephone number for the purpose of being contacted by the lay health worker
* NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Patient and clinician participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. This protocol does not permit use of Legally Authorized Representative NOTE: For this study, in the OPEN registration, clinician participants will be listed as their own treating investigator. However, clinician participants must not consent themselves or sign their own eligibility criteria forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2026-05-03 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-07-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with any hospitalization | Within 12 months of enrollment
  The primary analysis will be conducted using multivariable logistic regression, adjusting for stratification factors as covariates.

SECONDARY OUTCOMES:
Proportion of patients with 0 versus >= 1 of the combined endpoint of hospitalizations or emergency room (ER) visits | Up to 12 months
  Logistic, linear, and negative binomial regression models will be used, as appropriate for the given endpoint. Each regression analysis will include covariate adjustment for the stratification variables.
Number of hospitalizations as a continuous outcome | Up to 12 months
  Logistic, linear, and negative binomial regression models will be used, as appropriate for the given endpoint. Each regression analysis will include covariate adjustment for the stratification variables.
Number of hospitalizations or ER visits | Up to 12 months
  Logistic, linear, and negative binomial regression models will be used, as appropriate for the given endpoint. Each regression analysis will include covariate adjustment for the stratification variables.
Intensive end-of-life care | Up to 12 months
  Logistic, linear, and negative binomial regression models will be used, as appropriate for the given endpoint. Each regression analysis will include covariate adjustment for the stratification variables.
Anxiety | At 3 months after enrollment
  Logistic, linear, and negative binomial regression models will be used, as appropriate for the given endpoint. Each regression analysis will include covariate adjustment for the stratification variables. Baseline score will also be included as a model covariate.
Depression | At 3 months after enrollment
  Logistic, linear, and negative binomial regression models will be used, as appropriate for the given endpoint. Each regression analysis will include covariate adjustment for the stratification variables. Baseline score will also be included as a model covariate.

OTHER OUTCOMES:
Goals of care communication | Up to 12 months
  Abstracted from the electronic health record. Will assess differential impact by income and race and ethnicity.
Emergency room visits | Up to 12 months
  Will assess differential impact by income and race and ethnicity.
Patient-reported anxiety | At baseline, 3 months, and 6 months
  Measured using Patient Reported Outcomes Measurement Information System (PROMIS) version 1.0 Short Form Anxiety. Will assess differential impact by income and race and ethnicity.
Patient-reported depression | At baseline, 3 months, and 6 months
  Measured using PROMIS version 1.0 Short Form Depression. Will assess differential impact by income and race and ethnicity.
Patient-reported quality of communication with clinical staff | At baseline, 3 months, and 6 months
  Assessed using the Heard and Understood questionnaire. Will assess differential impact by income and race and ethnicity.
Patient-reported experiences with end of life care discussions | At baseline, 3 months, and 6 months
  Will be measured using the Prognostic Awareness and Treatment Preferences instrument. Will assess differential impact by income and race and ethnicity.
Hospitalizations alone | Up to 12 months
  Will be evaluated as time-to-event analysis. Will assess differential impact by income and race and ethnicity.
Hospitalizations and ER visits | Up to 12 months
  Will be evaluated as time-to-event analysis. Will assess differential impact by income and race and ethnicity.
ER visits | Up to 12 months
  Will be evaluated as time-to-event analysis. Will assess differential impact by income and race and ethnicity.
Percentage of approached sites that can map the electronic health record query (Feasibility) | Up to 6 years
  Feasibility goal for this implementation outcome is >= 90%.
Percentage of sites that can run the machine learning (ML) algorithm Python code on site (Feasibility) | Up to 6 years
  Feasibility goal for this implementation outcome is >= 90%.
Percentage of sites where ML retraining is not necessary prior to trial activation (Feasibility) | Up to 6 years
  Feasibility goal for this implementation outcome is >= 50%.
Percentage of eligible patients who consent to study (Adoption) | Up to 6 years
  Adoption goal for this implementation outcome is >= 50%.
Percentage of patients enrolled in the intervention arm who engage with the lay health workers at least once a month for first 6 months, prior to death, or prior to transition to hospice (Fidelity) | Up to 6 years
Acceptability of intervention | At 6 months after trial enrollment
  Assessed during mixed-methods interviews among intervention participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi B Parikh, Principal Investigator — SWOG Cancer Research Network